CLINICAL TRIAL: NCT02317575
Title: Safety, Tolerability, Pharmacokinetics and Glucodynamics of Multiple Insulin Lispro (LY900014) Formulations
Brief Title: A Study of LY900014 Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15645; I8B-FW-ITRA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2015-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: LY900014 Test A (Experimental): Test Formulation A. Single dose of LY900014 administered subcutaneously (SC) in one of five periods.
  Interventions: Biological: LY900014
- Part A:Insulin Lispro (Experimental): Reference formulation. 15 U insulin lispro administered SC in one of five periods.
  Interventions: Biological: Insulin Lispro
- Part A: LY900014 Test B (Experimental): Test Formulation B. Single dose LY900014 administered subcutaneously (SC) in one of five periods.
  Interventions: Biological: LY900014
- Part A: LY900014 Test C (Experimental): Test Formulation C. Single dose LY900014administered subcutaneously (SC) in one of five periods.
  Interventions: Biological: LY900014
- Part A: LY900014 Test D (Experimental): Test Formulation D. Single dose LY900014administered subcutaneously (SC) in one of five periods.
  Interventions: Biological: LY900014
- Part B: LY900014 (Experimental): Test formulation selected from Part A. Single dose of LY900014 administered SC in one of four periods.
  Interventions: Biological: LY900014

INTERVENTIONS:
Biological: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: Part A: LY900014 Test A; Part A: LY900014 Test B; Part A: LY900014 Test C; Part A: LY900014 Test D; Part B: LY900014
Biological: Insulin Lispro — Administered SC
  Other Names: LY275585
  Arms: Part A:Insulin Lispro

SUMMARY:
This study evaluated four test formulations of a glucose lowering drug (LY900014) administered by injection under the skin of the abdomen. The study was conducted in healthy people to investigate how the human body handles LY900014 and the effect of LY900014 on blood sugar levels. Side effects and tolerability were documented. The study was to be conducted in two parts (Part A and Part B) to achieve its objectives. Each part of the study was to last for about 11 to 12 weeks, including screening and follow up. Screening was required within 28 days prior to entering into either study Part A or Part B. Part B was not executed because no suitable formulation was identified.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female (not pregnant and agreeable to take birth control measures until one month after study completion)
* Have a body mass index (BMI) of 18.5 to 30 kilogram per square meter (kg/m^2), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Are nonsmokers, have not smoked for at least 2 months prior to entering the study, and agree not to smoke (cigars, cigarettes, or pipes) or use smokeless tobacco for the duration of the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days from a clinical trial or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part B was not executed and no data were collected.
Pre-assignment Details: Part A was a 5-period crossover study of four LY900014 formulations (Tests A, B, C, and D) and insulin lispro (Reference (R)). A minimum of 3 days washout between each period.
Groups:
- Part A Sequence 1, CDABR: Period 1: LY900014 Test C, Period 2: LY900014 Test D, Period 3: LY900014 Test A, Period 4: LY900014 Test B, Period 5: Reference (R) = insulin lispro
- Part A Sequence 2, ABDRC: Period 1: LY900014 Test A, Period 2: LY900014 Test B, Period 3: LY900014 Test D, Period 4: Reference (R) = insulin lispro, Period 5: LY900014 Test C
- Part A Sequence 3, BCRAD: Period 1: LY900014 Test B, Period 2: LY900014 Test C, Period 3: Reference (R) = insulin lispro, Period 4: LY900014 Test A, Period 5: LY900014 Test D
- Part A Sequence 4, DRBCA: Period 1: LY900014 Test D, Period 2: Reference (R) = insulin lispro, Period 3: LY900014 Test B, Period 4: LY900014 Test C, Period 5: LY900014 Test A
- Part A Sequence 5, RACDB: Period 1: Reference (R) = insulin lispro, Period 2: LY900014 Test A, Period 3: LY900014 Test C, Period 4: LY900014 Test D, Period 5: LY900014 Test B
Period: Period 1
Arm/Group | Part A Sequence 1, CDABR | Part A Sequence 2, ABDRC | Part A Sequence 3, BCRAD | Part A Sequence 4, DRBCA | Part A Sequence 5, RACDB
Started | 5 | 6 | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 5 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 6 | 6 | 6
Not Completed | 1 | 1 | 0 | 0 | 0
Not completed — Difficulty with venous cannulation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part A Sequence 1, CDABR | Part A Sequence 2, ABDRC | Part A Sequence 3, BCRAD | Part A Sequence 4, DRBCA | Part A Sequence 5, RACDB
Started | 4 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A Sequence 1, CDABR | Part A Sequence 2, ABDRC | Part A Sequence 3, BCRAD | Part A Sequence 4, DRBCA | Part A Sequence 5, RACDB
Started | 4 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Part A Sequence 1, CDABR | Part A Sequence 2, ABDRC | Part A Sequence 3, BCRAD | Part A Sequence 4, DRBCA | Part A Sequence 5, RACDB
Started | 4 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Part A Sequence 1, CDABR | Part A Sequence 2, ABDRC | Part A Sequence 3, BCRAD | Part A Sequence 4, DRBCA | Part A Sequence 5, RACDB
Started | 4 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Overall Study: Participants were administered LY900014 SC Tests A, B, C, and D, with that of 15 U of insulin lispro alone (Reference) in healthy subjects.
Arm/Group | Overall Study
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 27
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 28
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 72.60 (9.07)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per meter squared (kg/m²)] | 24.43 (2.21)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Pharmacokinetics (PK ): Area Under the Concentration Curve From Zero to the Last Recorded Time Post Dose (AUC0-tlast)
Time Frame: 30 minutes predose, 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, and 300 minutes postdose
Population: All participants who received at least 1 dose of study drug and completed the dose sequence.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: picomol times hour per liter (pmol*h/L)
Groups:
- Part A: Formulation A, LY900014; Part A: Formulation B, LY900014; Part A: Formulation C, LY900014; Part A: Formulation D, LY900014: Single dose LY900014 administered subcutaneously (SC) in one of five periods
- Part A: Reference: 15 U of insulin lispro administered subcutaneously (SC) in one of five periods
Arm/Group | Part A: Formulation A, LY900014 | Part A: Formulation B, LY900014 | Part A: Formulation C, LY900014 | Part A: Formulation D, LY900014 | Part A: Reference
Number analyzed (Participants) | 27 | 27 | 28 | 27 | 27
picomol times hour per liter (pmol*h/L) | 1720 (20) | 1740 (17) | 1810 (21) | 1750 (19) | 1690 (19)

2. Secondary Outcome: Part A: Visual Analog Scale (VAS) Score for Injection Site Pain
Description: The Visual Analog Scale (VAS) assessed injection site pain on a scale of 0-100 millimeter (mm) range (0 = no pain and 100 worst imaginable pain).
Time Frame: Predose, 1, 20, 60 minutes postdose and at the end of the clamp procedure
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Groups:
- Part A: Formulation A, LY900014; Part A: Formulation B, LY900014; Part A: Formulation D, LY900014: 15 U LY900014 administered SC in one of five periods
- Part A: Formulation C, LY900014: 115 U LY900014 administered SC in one of five periods
Arm/Group | Part A: Formulation A, LY900014 | Part A: Formulation B, LY900014 | Part A: Formulation C, LY900014 | Part A: Formulation D, LY900014 | Part A: Reference
Number analyzed (Participants) | 27 | 27 | 28 | 27 | 27
millimeter (mm)
  1 minute | 0.1 (0.6) | 2.1 (6.5) | 1.8 (4.8) | 1.3 (4.7) | 0.5 (1.9)
  20 minutes | 0 (0) | 0 (0) | 0 (0) | 2.0 (9.6) | 0 (0)
  60 minutes | 0 (0) | 0 (0) | 0 (0) | 1.1 (6.0) | 0 (0)
  End of clamp | 0 (0) | 0 (0) | 0 (0) | 0 (0.2) | 0 (0)

3. Secondary Outcome: Part A: Total Amount of Glucose Infused (Gtot) Over the Duration of Clamp
Description: Gtot is the total glucose infusion over the clamp duration and is used to measure the study drug action over time as measured by the euglycaemic clamp procedure.
Time Frame: Every 10 minutes for 30 minutes predose, every 2.5 minutes for 30 minutes, then every 5 minutes for 120 minutes, then every 10 minutes for 300 minutes postdose
Population: All participants who received at least 1 dose of study drug and completed the dose sequence.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: milligram (mg)
Groups:
- Part A: Formulation C, LY900014; Part A: Formulation D, LY900014: 15 U LY900014 administered SC in one of five periods
Arm/Group | Part A: Formulation A, LY900014 | Part A: Formulation B, LY900014 | Part A: Formulation C, LY900014 | Part A: Formulation D, LY900014 | Part A: Reference
Number analyzed (Participants) | 27 | 27 | 28 | 27 | 27
milligram (mg) | 78372 (29) | 81776 (41) | 82365 (35) | 80186 (34) | 75571 (37)

4. Secondary Outcome: Part B: Total Amount of Glucose Infused (Gtot) Over the Duration of the Clamp - Interparticipant Variability
Description: as for outcome 3
Time Frame: Every 10 minutes for 30 minutes predose, every 2.5 minutes for 30 minutes, then every 5 minutes for 120 minutes, then every 10 minutes for 300 minutes, then every 20 minutes from 300 to 480 minutes postdose
Population: Zero participants were analyzed as Part B was not executed.
Groups:
- Part B:LY900014: Formulation selected from Part A. Single dose of LY900014 administered SC in one of four periods.
Arm/Group | Part B:LY900014
Number analyzed (Participants) | 0

5. Secondary Outcome: Part B: Pharmacokinetics (PK): Area Under the Concentration Curve From Zero to the Last Recorded Time Post Dose (AUC0-tlast) - Interparticipant Variability
Time Frame: Predose, 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, and 300 minutes postdose
Population: Zero participants were analyzed as Part B was not executed.
Arm/Group | Part B:LY900014
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Part A: Forumulation C, LY900014; Part A: Forumulation D, LY900014: Single dose LY900014 administered subcutaneously (SC) in one of five periods
- Part A: Reference: 15 U insulin lispro administered subcutaneously (SC)
Arm/Group | Part A: Formulation A, LY900014 | Part A: Formulation B, LY900014 | Part A: Forumulation C, LY900014 | Part A: Forumulation D, LY900014 | Part A: Reference
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/28 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 5/27 | 5/27 | 2/28 | 6/27 | 2/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Formulation A, LY900014 (N=27) | Part A: Formulation B, LY900014 (N=27) | Part A: Forumulation C, LY900014 (N=28) | Part A: Forumulation D, LY900014 (N=27) | Part A: Reference (N=27)
Catheter site related reaction (General disorders) | 5 (5) | 5 (5) | 2 (2) | 6 (6) | 2 (2)

LIMITATIONS AND CAVEATS:
Part B was not executed per protocol because no formulation was identified in Part A.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days